CLINICAL TRIAL: NCT06343688
Title: Examination of the Instant Effect of DAFO Use on Balance and Lower Extremity Gross Motor Functions in Individuals With Spastic Diplegic Cerebral Palsy
Brief Title: "Immediate Effect of DAFO on Gross Motor Function and Balance in Diplegic Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Principal Investigator, Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-5
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Diplegic Cerebral Palsy
Keywords: cerebral palsy; Diplegia; Spastic; orthosis; balance
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Group: "The Gross Motor Function Classification System (GMFCS) will be used to classify children's gross motor levels, the Manual Abilities Classification System (MACS) for hand skills, the Communication Function Classification System (CFCS) for communication skills, and the Eating and Drinking Ability Classification System (EDACS) for feeding skills. Additionally, the Gross Motor Function Measure (GMFM-88) items D and E will be used to assess motor skills, the Wii Balance Board for testing balance, the Pediatric Berg Balance Scale, and the functional reach test will be utilized. The balance and gross motor functions of the included children will be evaluated in two different ways: with and without DAFO."
  Interventions: Other: "Assessment of Balance and Lower Extremity Gross Motor Function with and without DAFO"

INTERVENTIONS:
Other: "Assessment of Balance and Lower Extremity Gross Motor Function with and without DAFO" — "Measurements will be conducted with the child's custom-made DAFO (Dynamic Ankle-Foot Orthosis) and barefoot."

SUMMARY:
" Study will investigate the immediate effect of DAFO usage on balance and gross motor functions in individuals with spastic diplegic cerebral palsy. The study is planned to be conducted with children aged 4-15 who have GMFCS levels 1 and 2 and who are willing to participate along with their families at the Turkey Spastic Children Foundation Metin Sabancı Special Education and Rehabilitation Center. During the dates of the study, children who meet the inclusion criteria will be evaluated. Demographic information such as age, height, and weight will be obtained for the participating children. To classify the gross motor levels of the children, the Gross Motor Function Classification System (GMFCS), the Manual Abilities Classification System (MACS) for hand skills, the Communication Function Classification System (CFCS) for communication skills, and the Eating and Drinking Ability Classification System (EDACS) for feeding skills will be used. In addition, the Gross Motor Function Measure (GMFM-88) items D and E for assessing motor skills, the Wii Balance Board for testing balance, the Pediatric Berg Balance Scale, and the functional reach test will be utilized. The balance and gross motor functions of the included children will be assessed in two different ways: with and without DAFO. Data analysis will be conducted by a blinded statistician who is not part of the research team. IBM SPSS 26 (Statistical Package for Social Sciences) will be used for statistical analysis of the data. Normality of continuous variables will be assessed using the Kolmogorov-Smirnov test. If continuous variables follow a normal (parametric) distribution, paired sample t-tests will be conducted on pre-test and post-test data. If the data are non-parametric, Wilcoxon test will be used. Pearson chi-square test or Spearman correlation coefficient will be used to determine the relationship between variables based on assumptions. Results will be evaluated at a significance level of p < 0.05 with a 95% confidence interval."

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a group of motor disorders resulting from non-progressive damage to the immature brain, leading to movement and posture impairments. Approximately 2 to 3 out of every 1000 children worldwide are born with CP. Prevalence studies conducted before 1990 reported an increasing trend in CP prevalence. However, prevalence is not static, and improvements in prenatal care due to advancements in healthcare have led to a slight decrease in prevalence. A study in 2013 reported a prevalence rate between 2.2% and 2.3%.

Children with CP exhibit various symptoms such as contractures, spasticity, and coordination disorders, mainly affecting the musculoskeletal and nervous systems. These symptoms adversely affect their mobility, functional abilities, and quality of life.

CP is classified into three types based on movement disorder: spastic, dyskinetic, and ataxic, and into four classes based on the pattern of involvement: quadriplegic, hemiplegic, diplegic, and monoplegic. Among these, diplegic CP is the most common type, accounting for 30-35% of cases. Diplegic CP primarily affects the lower extremities more than the upper extremities. Children with diplegic CP often exhibit a pathological gait characterized by pes equinovarus, genu valgus, excessive knee flexion, increased hip adduction, and internal rotation.

The management of CP involves physiotherapy, orthotic support, surgeries, temporary medical interventions, and speech-language therapy. Orthoses, such as Ankle-Foot Orthoses (AFOs), are commonly used in CP rehabilitation. Dynamic Ankle-Foot Orthoses (DAFOs) have emerged as a popular alternative to AFOs in diplegic CP. DAFOs are designed to control muscle tone and prevent foot deformities by providing proper support to the foot's plantar surface. They allow for partial movement due to their flexible and thinner structure compared to rigid AFOs.

Studies have shown that DAFOs significantly impact gross motor skills in children with CP. DAFOs aim to manage foot deformities, increase support, facilitate skill training, and improve mobility during standing and walking.

1. Examine the effect of DAFO use on balance in children with diplegic CP.
2. Investigate the effect of DAFO use on lower extremity gross motor functions in children with diplegic CP.
3. Explore the impact of DAFO use on functionality in children with diplegic CP.

Upon obtaining meaningful results, this study aims to contribute to clinical practice and scientific research in the field of CP rehabilitation.

**Materials and Methods / Design**

**Sample Size:** The sample size of this study was determined based on a power analysis conducted using data from a similar study. With a significance level (α) of 0.05, power (1- β) of 0.90, and effect size (Cohen's d) of 0.97, it was calculated that a total of 38 patients would be sufficient to detect the difference. However, considering possible withdrawals or issues with completing the analysis, the sample size was set at a minimum of 40.

**Procedure:** The study will be conducted with the participation of children aged 4-15 diagnosed with cerebral palsy (CP) at levels 1 and 2 according to the Gross Motor Function Classification System (GMFCS) at the Metin Sabancı Special Education and Rehabilitation Center for Children with Spastic Disabilities in Turkey. The evaluation will take place among children who meet the predefined inclusion criteria during the specified dates.

Demographic information such as age, height, and weight will be collected for the participating children. Classification systems such as the Gross Motor Function Classification System (GMFCS) for assessing gross motor function, the Manual Ability Classification System (MACS) for assessing manual abilities, the Communication Function Classification System (CFCS) for assessing communication abilities, and the Eating and Drinking Ability Classification System (EDACS) for assessing eating and drinking abilities will be used. Additionally, the Gross Motor Function Measure (GMFM), Pediatric Balance Scale (PBS), and functional reach test will be employed to evaluate motor skills and balance. The children's balance and gross motor functions will be assessed using different evaluation methods with and without the use of Dynamic Ankle Foot Orthoses (DAFOs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Spastic Diplegic type of cerebral palsy
* Age between 4 and 15 years
* Using bilateral Dynamic Ankle-Foot Orthosis (DAFO)
* Communication Function Classification System (CFCS) level between 1 and 2
* Gross Motor Function Classification System (GMFCS) level between 1 and 2
* Willingness to participate in the study

Exclusion Criteria:

* Having experienced lower extremity fractures or muscle-tendon and bone surgery in the past 6 months, or having undergone spinal or orthopedic surgery affecting the lower extremities
* Exposure to any pharmacological agent or intervention inhibiting spasticity in the past 6 months.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with spastic diplegic cerebral palsy who are independently walking and aged between 4 and 15 years.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Wii Balance Board | day 1
  The Wii Balance Board transmits vertical ground reaction forces from four corners of the device to the Wii system via Bluetooth when an individual stands on it. The Fizyosoft Balance System, developed by engineers and physiotherapists, will be used to assess static balance in participating children. Swing speeds measured using the Wii Balance Board, which establishes a Bluetooth connection with a computer, will be indexed. The dimensions of the Wii Balance Board are approximately 45 x 26.5 cm, with a weight capacity of approximately 150 kg. Children will be instructed to stand on the device with their feet parallel to each other and remain motionless for 15 seconds, with measurements taken with eyes open and closed. The coordinates of the individuals' center of pressure (COPx, COPy) will be recorded in centimeters (cm), while the performance value will be recorded as a percentage in the system.""A high deviation from the x and y coordinates indicates poor balance."
"The Gross Motor Function Measure-88 (D-E) (GMFM-88) | day 1
  To assess changes in lower extremity gross motor function in children with cerebral palsy, the D (Standing) and E (Walking/Running/Jumping) sections of the GMFM-88 test will be used. The D section consists of 12 questions ranging from 52 to 64, and the E section consists of 23 questions ranging from 65 to 88. A total of 35 questions will be evaluated""Low scores indicate poor gross motor function."
The Functional Reach Test | day 1
  The Functional Reach Test is a dynamic balance assessment method. It measures the maximum distance that can be reached forward and sideways while standing upright. The reached distance is calculated as the difference between the maximum distance reached while standing upright without lifting the heels from the ground and the maximum distance reached while maintaining hip flexion without lifting the heels from the ground. This method, commonly used in adults, is employed to evaluate the ability to maintain balance and stability. Studies have shown that this test, designed for adults, can also be applied to children.Low scores indicate poor balance.
"The Pediatric Berg Balance Scale (PBBS) | day 1
  The Pediatric Berg Balance Scale (PBBS) is a test consisting of 14 questions related to parameters such as standing up from sitting, standing, transfers, walking, turning, etc. Each question is scored from 0 to 4, and the time taken to perform the desired activity is recorded. At the end of the test, the total score obtained by the individual is calculated and recorded. Validity and reliability studies of this scale have been conducted for various neurological diseases such as Parkinson's disease, stroke, spinal cord injuries, etc., as well as for geriatrics.""Higher scores indicate better balance levels."

SECONDARY OUTCOMES:
"The Eating and Drinking Ability Classification System (EDACS) | day 1
  It classifies eating and drinking abilities of children with cerebral palsy from the age of 3 onwards. EDACS defines an individual's eating and drinking abilities at 5 different skill levels, focusing on activities such as sucking, biting, chewing, swallowing, and holding food or liquid in the mouth. Level I signifies the least impact for children with cerebral palsy, while Level V indicates severe impact. It categorizes all aspects of eating and drinking performance, including both motor and sensory components. The system provides a broad distinction between different levels of functional ability. EDACS is not a scale that assesses components of eating and drinking in detail. Changes in eating and drinking performance occur due to growth, physical development, and experience. The child will be classified into one of the levels ranging from 1 to 5.""In the scale, a high score indicates a significant impact and poor functioning of the child."
"The Manual Abilities Classification System (MACS) | day 1
  The Manual Abilities Classification System (MACS) is a scale designed to determine how children with cerebral palsy aged 4-18 use their hands to hold objects during daily activities. Classified into 5 levels, MACS is based on the child's ability to grasp objects independently and the need for assistance and adaptation in performing hand-related activities in daily life. Level I signifies the least impact for children with cerebral palsy, while Level V indicates severe impact. To understand how the child holds objects in daily life, information should be obtained from those who spend the most time with the child. MACS is a classification system aimed at reflecting the overall condition of hand use in daily life, rather than the child's best performance during an activity. The child will be classified into one of the levels ranging from 1 to 5.""In the scale, a high score indicates a significant impact and poor functioning of the child."
"The Gross Motor Function Classification System (GMFCS) | day 1
  GMFCS utilizes gross motor skills such as head control, mobilization, transfer activities, walking and running, jumping, and navigating on uneven or non-level surfaces to define a child's level of ability. GMFCS categorizes children based on how they routinely ambulate in home, school, or community settings and according to common criteria. Level I signifies the least impact for children with cerebral palsy, while Level V indicates severe impact. This system was expanded in 2007 to include age ranges of 12-15 and 15-18, emphasizing concepts specific to the World Health Organization's international classification of functioning, disability, and health. The child will be classified into one of the levels ranging from 1 to 5.""In the scale, a high score indicates a significant impact and poor functioning of the child."
"The Communication Function Classification System (CFCS) | day 1
  CFCS Levels:
  Level I: Effective sender and receiver with familiar and unfamiliar partners Level II: Effective but slow sender and receiver with familiar and/or unfamiliar partners Level III: Effective sender and receiver with familiar partners Level IV: Inconsistent sender and/or receiver with familiar partners Level V: Rarely effective sender and receiver even with familiar partners
  The child will be classified into one of the levels ranging from 1 to 5.""In the scale, a high score indicates a significant impact and poor functioning of the child."

CONTACTS AND LOCATIONS:
Overall Officials: özge karanlık, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided